CLINICAL TRIAL: NCT01230645
Title: A Randomized, Single-blind, Placebo-controlled, Parallel Group Study to Investigate the Effects of Intranasal RV568 (400μg) Administered Twice Daily to Adult Male Volunteers Experimentally Inoculated With Live Respiratory Syncytial Virus
Brief Title: RV568 - Viral Challenge With RSV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Respivert Ltd (Industry)
Responsible Party: Dr Garth Rapeport, Respivert Ltd
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RVH003; 2010-021527-26 (EudraCT Number)
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- RV568 treatment group (Experimental)
  Interventions: Drug: RV568
- Placebo treatment group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RV568 — RV568 400 ug administered as nasal drops twice daily for 10 days (Day -1 to Day 8)
  Arms: RV568 treatment group
Drug: Placebo — Placebo administered as nasal drops twice daily for 10 days (Day -1 to Day 8)
  Arms: Placebo treatment group

SUMMARY:
RV568 is being developed for the treatment of diseases such as asthma, COPD and allergic rhinitis (e.g. hayfever). The main aim of this study is to investigate whether RV568 is effective in reducing the inflammation caused by viral infections such as RSV (respiratory syncytial virus).

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects aged 18 - 45 years
* agreeable to use adequate contraception throughout the study
* negative hepatitis B, hepatitis C and HIV screen
* negative drugs of abuse, alcohol and nicotine screen
* able to provide written informed consent and be willing to comply with the study restrictions and requirements
* low titres of RSV neutralising antibody measured during screening

Exclusion Criteria:

* acute or chronic illness or clinically relevant abnormality noted at the screening visit
* presence of febrile illness or symptoms of upper or lower respiratory tract infection in the 28 days prior to viral inoculation
* history of asthma, COPD, pulmonary hypertension, reactive airway disease, or any chronic lung condition
* diabetes
* history or evidence of autoimmune disease or known impaired immune responsiveness
* recent (within the last 3 years) and/or recurrent history of autonomic dysfunction
* anatomic or neurological abnormality impairing the gag reflex or associated with an increased risk of aspiration, any abnormality significantly altering the anatomy of the nose or nasopharynx. Known IgA deficiency, immotile cilia syndrome, or Kartagener's syndrome. Any nasal or sinus surgery within 4 months prior to virus administration.
* history of smoking in the past 6 months
* positive test for drugs or alcohol at screening
* inadequate venous access
* abnormal pulmonary function at screening
* abnormal laboratory or ECG at screening
* acute or chronic use of medication to treat nasal congestion
* use of any prescription drugs, herbal supplements, within 4 weeks prior to virus challenge, and/or over-the-counter medication, dietary supplements within 2 weeks prior to virus challenge
* treatment with systemic glucocorticoids, antiviral drugs, immunoglobulins or blood transfusions within 1 month, or any other cytotoxic or immunosuppressive drug within 6 months prior to dosing. Receipt of any systemic chemotherapy agent at any time
* treatment with any investigational drug within 3 months, or prior participation in a clinical trial of any RSV IMP, medication or experimental RSV viral challenge delivered directly to the respiratory tract within 1 year prior to dosing, or receipt of more than 4 investigational drug within 12 months
* history of multiple and recurring allergies and/or adverse reaction to any components of the challenge virus preparation
* allergy to gentamicin
* significant history of seasonal hay fever or seasonal allergic rhinitis (SAR), perennial allergic rhinitis (PAR), or chronic nasal or sinus condition
* intention to travel between first and last visit (to countries for which vaccinations are recommended or where high risk of infection exists)
* healthcare workers (including doctors, nurses, medical students and allied healthcare professionals) anticipated to have patient contact within two weeks of viral challenge
* household member or close contact (for an additional 2 weeks after discharge from the isolation facility) who is:

  1. less than 3 years of age;
  2. any person with any known immunodeficiency;
  3. any person receiving immunosuppressant medications;
  4. any person undergoing or soon to undergo cancer chemotherapy within 28 days of viral challenge;
  5. any person who has diagnosed emphysema or COPD, is elderly residing in a nursing home, or with severe lung disease or medical condition including but not exclusive to the conditions listed below; or
  6. any person who has received a transplant (bone marrow or solid organ)
* employees or relatives of Retroscreen Virology or RespiVert Ltd
* other finding in the medical interview, physical exam, or screening investigations that, in the opinion of the Investigator, deem the subject unsuitable for the study
* subjects who in the opinion of their general practitioner or the Investigator, should not participate in the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
IL8 induction in nasal wash samples | 16 day quarantine period

SECONDARY OUTCOMES:
RSV viral load | 16 day quarantine period
Changes in symptoms of RSV infection | 16 day quarantine period
Assessment of mucus weight and tissue counts | 16 day quarantine period
Viable nasal cell counts in nasal washes | 16 day quarantine period
Frequency of RSV infection | 16 day quarantine period
Plasma RV568 levels | 16 day quarantine period
Assessment of IL6 in nasal wash samples | 16 day quarantine period

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Gilbert, MD, Principal Investigator — Retroscreen Virology Ltd.
Locations (1):
- Retroscreen Virology Ltd, London, United Kingdom